CLINICAL TRIAL: NCT06477471
Title: A Preliminary Investigation of the Safety and Effectiveness of Oral Probiotics Supplementation for Reducing the Risk of Kidney Stone in Adults With Recurrent Kidney Stone Colic or Acute Episode of Colicky Pain: An Open-Label, Single-Arm, Prospective, Interventional, Proof-of-Science Study
Brief Title: A Clinical Study to Determine the Safety and Efficacy of An Oral Probiotic. Supplementation in Reducing the Risk of Kidney Stone in Adults With Recurrent Kidney Stone Colic or Acute Episode of Colicky Pain.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NovoBliss Research Pvt Ltd (Other)
Collaborators: Meteoric Biopharmaceuticals Pvt. Ltd. (Industry)
Responsible Party: Principal Investigator, Dr Nayan Patel, Principal Investigator- Medical Director, NovoBliss Research Pvt Ltd
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NB240020-MB
Record Dates: First submitted 2024-06-07; First posted 2024-06-27 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Recurrent Kidney Stones With Colicky Pain

STUDY DESIGN:
Intervention Model Description: An Open-Label, Single-Arm, Prospective, Interventional, Proof-of-Science Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Recurrent Kidney Stone with Colicky Pain (Experimental): Take one slow-release capsule twice a day, after meal, orally.
  Interventions: Other: MetProrenes

INTERVENTIONS:
Other: MetProrenes — Take one slow-release capsule twice a day, after meal.

SUMMARY:
A Preliminary Investigation of the Safety and Effectiveness of Oral Probiotics Supplementation for Reducing the Risk of Kidney Stone in Adults with Recurrent Kidney Stone Colic or Acute Episode of Colicky Pain: An Open-Label, Single-Arm, Prospective, Interventional, Proof-of-Science Study.

14 adults, with recurrent kidney stone colic or acute episode of colicky pain will be enrolled to ensure 12 subjects complete the study

DETAILED DESCRIPTION:
Potential subjects will undergo screening based on predefined inclusion and exclusion criteria only after obtaining written informed consent.

Subjects shall be instructed to visit the facility for the following scheduled visits:

* Visit 01 [Day 01]: Screening, baseline evaluations, enrolment and test treatment dispensing.
* Visit 02 [Day 14 (± 2 days)]: Treatment End, Follow-up Evaluations.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is an adult aged between 18 to 55 years old.
2. The subject has a history of recurrent kidney stone colic or acute episode of colicky pain on clinical examination by Physician.
3. Subject having refrigerator at their home for storage of test product.
4. The subject is willing to provide written informed consent and comply with study procedures, including overnight stay for 24 hours at the study centre during both visits.
5. The subject is willing to abide by the study protocol and restrictions, including abstaining from using any other oral or topical treatments for kidney stone colic during the study period.
6. The subject is in a stable medical condition, not requiring immediate intervention or hospitalization.
7. If the subject is female, she is willing to use a highly effective method of contraception throughout the clinical investigation.

   1. Females of childbearing potential must practice and maintain an established method of birth control (e.g., IUD, hormonal implant device/injection, birth control pills, diaphragm, condoms with spermicide, partner vasectomy, or abstinence).
   2. Non-childbearing potential females who are surgically sterile, post-menopausal for at least 1 year, or have had a tubal ligation, must have been using hormonal contraception for at least 6 months and agree to continue using the same contraception for the study duration.

Exclusion Criteria:

1. The subject has a history of severe renal impairment or chronic kidney disease.
2. The subject is pregnant/lactating, or is planning on become pregnant during the course of the study.
3. The subject has presence of significant medical or psychiatric conditions that may interfere with study participation or interpretation of results.
4. The subject has a history of substance abuse or dependence.
5. The subject has severe systemic complications of viral infections, cardiovascular disorders, neurological disorders, renal disorders, or autoimmune disorders.
6. The subject has participated in clinical studies or received any investigational agent in the previous 30 days.
7. The subject has any condition that, in the investigator's judgment, would compromise the subject's safety or study integrity.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Estimated)
Dates: Start 2024-07-30 (Estimated); Primary Completion 2024-08-13 (Estimated); Study Completion 2024-08-13 (Estimated)

PRIMARY OUTCOMES:
Change in the colicky pain | On Day 01 (before administration) for baseline, and post-dosage on Day 14 (±2 days).
  Evaluate the effect of the test treatment in term of change in the colicky pain determined using the VAS scoring where 0 indicates no pain and 10 indicates severe pain
Changes in Urine Calcium | On Day 01 (before administration) for baseline, and post-dosage on Day 14 (±2 days).
  Assessment of the effectiveness of the test treatment in terms of changes in Urine Calcium examined by urinalysis after 24h-urine collection
Changes in Urine Sodium | On Day 01 (before administration) for baseline, and post-dosage on Day 14 (±2 days).
  Assessment of the effectiveness of the test treatment in terms of changes in Urine Sodium examined by urinalysis after 24h-urine collection
Changes in Urine Oxalate | On Day 01 (before administration) for baseline, and post-dosage on Day 14 (±2 days).
  Assessment of the effectiveness of the test treatment in terms of changes in Urine Oxalate examined by urinalysis after 24h-urine collection
Changes in Urine pH | On Day 01 (before administration) for baseline, and post-dosage on Day 14 (±2 days).
  Assessment of the effectiveness of the test treatment in terms of changes in Urine pH examined by urinalysis after 24h-urine collection
Changes in Urine R/M | On Day 01 (before administration) for baseline, and post-dosage on Day 14 (±2 days).
  Assessment of the effectiveness of the test treatment in terms of changes in Urine R/M examined by urinalysis after 24h-urine collection

SECONDARY OUTCOMES:
Changes in Haemoglobin | On Day 01 (before administration) for baseline, and post-dosage on Day 14 (±2 days).
  Assessment of the safety of the test treatment in terms of abnormal changes in Haemoglobin
Changes in Haematocrit | On Day 01 (before administration) for baseline, and post-dosage on Day 14 (±2 days).
  Assessment of the safety of the test treatment in terms of abnormal changes in Haematocrit.
Changes in Red Blood count | On Day 01 (before administration) for baseline, and post-dosage on Day 14 (±2 days).
  Assessment of the safety of the test treatment in terms of abnormal changes in Red Blood Count.
Changes in Packed Cell Volume | On Day 01 (before administration) for baseline, and post-dosage on Day 14 (±2 days).
  Assessment of the safety of the test treatment in terms of abnormal changes in Packed cell volume Count.
Changes in Red Blood count morphology | On Day 01 (before administration) for baseline, and post-dosage on Day 14 (±2 days).
  Assessment of the safety of the test treatment in terms of abnormal changes in Red Blood Count morphology.
Changes in Mean corpuscular volume | On Day 01 (before administration) for baseline, and post-dosage on Day 14 (±2 days).
  Assessment of the safety of the test treatment in terms of abnormal changes in Mean corpuscular volume
Changes in mean corpuscular hemoglobin | On Day 01 (before administration) for baseline, and post-dosage on Day 14 (±2 days).
  Assessment of the safety of the test treatment in terms of abnormal changes in mean corpuscular hemoglobin
Changes in mean corpuscular hemoglobin concentration | On Day 01 (before administration) for baseline, and post-dosage on Day 14 (±2 days).
  Assessment of the safety of the test treatment in terms of abnormal changes in mean corpuscular hemoglobin concentration
Changes in red blood cell distribution width | On Day 01 (before administration) for baseline, and post-dosage on Day 14 (±2 days).
  Assessment of the safety of the test treatment in terms of abnormal changes in red blood cell distribution width
Changes in Total WBC count | On Day 01 (before administration) for baseline, and post-dosage on Day 14 (±2 days).
  Assessment of the safety of the test treatment in terms of abnormal changes in Total WBC count.
Changes in Differential WBC count | On Day 01 (before administration) for baseline, and post-dosage on Day 14 (±2 days).
  Assessment of the safety of the test treatment in terms of abnormal changes in Differential WBC count.
Changes in Platelet count | On Day 01 (before administration) for baseline, and post-dosage on Day 14 (±2 days).
  Assessment of the safety of the test treatment in terms of abnormal changes in Platelet count.
Changes in mean platelet volume | On Day 01 (before administration) for baseline, and post-dosage on Day 14 (±2 days).
  Assessment of the safety of the test treatment in terms of abnormal changes in mean platelet volume.
Changes in Plateletcrit | On Day 01 (before administration) for baseline, and post-dosage on Day 14 (±2 days).
  Assessment of the safety of the test treatment in terms of abnormal changes in Plateletcrit.
Changes in platelet distribution width | On Day 01 (before administration) for baseline, and post-dosage on Day 14 (±2 days).
  Assessment of the safety of the test treatment in terms of abnormal changes in platelet distribution width.
Changes inSerum Creatinine | On Day 01 (before administration) for baseline, and post-dosage on Day 14 (±2 days).
  Assessment of the safety of the test treatment in terms of abnormal changes in Serum Creatinine.
Changes in Serum Glutamic Pyruvic Transaminase | On Day 01 (before administration) for baseline, and post-dosage on Day 14 (±2 days).
  Assessment of the safety of the test treatment in terms of abnormal changes in Serum Glutamic Pyruvic Transaminase
Changes in Serum Glutamic-Oxaloacetic Transaminase | On Day 01 (before administration) for baseline, and post-dosage on Day 14 (±2 days).
  Assessment of the safety of the test treatment in terms of abnormal changes in Serum Glutamic-Oxaloacetic Transaminase

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Nayan K Patel, Principal Investigator — NovoBliss Research Pvt Ltd

IPD SHARING:
Plan to Share IPD: No